CLINICAL TRIAL: NCT03277482
Title: A Phase 1 Study of Durvalumab, Tremelimumab and Radiotherapy in Recurrent Gynecologic Cancer
Brief Title: Durvalumab, Tremelimumab + Radiotherapy in Gynecologic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Expansion cohort was not open
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Martin King, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-382
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Gynecological Cancer; Metastatic Cervical Cancer; Metastatic Ovarian Cancer; Metastatic Vaginal Cancer; Metastatic Vulvar Cancer; Metastatic Endometrial Cancer; Recurrent Cervical Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Vaginal Cancer; Recurrent Vulvar Cancer; Recurrent Endometrial Cancer
Keywords: Recurrent gynecological cancer; Metastatic Cervical Cancer; Metastatic Ovarian Cancer; Metastatic Vaginal Cancer; Metastatic Vulvar Cancer; Metastatic Endometrial Cancer; Recurrent Cervical Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Vaginal Cancer; Recurrent Vulvar Cancer; Recurrent Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Endometrial Neoplasms | interventions — durvalumab; tremelimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Phase I Safety Lead-In (Experimental): A modified 3+3 design will be used in this trial Lead-in phase with Durvalumab* and radiation therapy
  *q4 weeks durvalumab for 13 cycles or until progression
  Interventions: Drug: Durvalumab; Radiation: Radiation Therapy
- Phase I Radiation Dose Evaluation (Experimental): * Durvalumab
  * Tremelimumab* -- Start radiation dose from safety lead-in (level 0 or level -1) *q4 weeks durvalumab / tremelimumab for 4 cycles and continue durvalumab for 13 cycles or until disease progression
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is given by intravenous infusion every 4 weeks for a maximum of 13 doses over 52 weeks. One cycle is defined as every 4 weeks. Each infusion will take approximately 1 hour.
  Other Names: Imfinizi; MEDI4736
Drug: Tremelimumab — Tremelimumab is given by intravenous infusion every 4 weeks for a maximum of 4 doses over 16 weeks. One cycle is defined as every 4 weeks. If receiving both durvalumab and tremelimumab for the first 4 cycles, they will be given on the same day. Each infusion will take approximately 1 hour
  Other Names: CP-675,206; CP-675
  Arms: Phase I Radiation Dose Evaluation
Radiation: Radiation Therapy — Radiation treatment will begin on the same day as the first immunotherapy infusion or on the following day. The radiation treatment course is either 1 day or 5 days.

SUMMARY:
This research study is evaluating the safety and effectiveness of 2 immunotherapy drugs in combination with radiation therapy as a possible treatment for recurrent or metastatic gynecologic cancer.

The names of the immunotherapy drugs involved in this study are:

* Durvalumab
* Tremelimumab

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug or drugs and also tries to define the appropriate dose and combination of the investigational drugs to use for further studies. "Investigational" means that the drugs are being studied but have not been approved by the FDA (the U.S. Food and Drug Administration).

In this study, the combination of durvalumab and tremelimumab is considered to be investigational and as such has not been approved for this or any cancer.

-- Durvalumab and tremelimumab are immunotherapy drugs that may stop cancer cells from growing by activating the immune system. The immune system is one of the body's natural defenses against the growth of cancer cells. AstraZeneca has evaluated the effectiveness and side effects of both durvalumab and tremelimumab individually for many cancer types, including lung, head and neck cancer, and melanoma. These types of immunotherapy drugs are also being studied in ovarian, endometrial and cervical cancer. In addition, AstraZeneca has studied the combination of durvalumab and tremelimumab in participants with lung and pancreatic cancers. Based on these studies, AstraZeneca has determined the dosing, schedule and expected side effects for the 2 study drugs when delivered together.

In women with recurrent or metastatic gynecologic cancer, radiation therapy is often used to help with symptoms, such as bleeding, pain or swelling. Clinical reports have shown that radiation treatment can increase the body's response to an immunotherapy drug against tumors both within and outside the radiation field. This study is the first in which the combination of durvalumab, tremelimumab and abdominal or pelvic radiation is given to humans. The investigators hope that this combination with radiation will lead to a better treatment response to the immunotherapy drugs.

The investigators will also look to see if participants whose tumors contain a particular genetic make-up have a better response to immunotherapy and radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Participants must have histologically or cytologically confirmed endometrial, ovarian (including ovarian epithelial, fallopian tube, primary peritoneal), cervical, vaginal, or vulvar cancer that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Participants must have measurable disease, defined as at least 1 lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥20 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease. See also 3.1.10 as all measurable/target lesions must not be located within the planned radiation field for the expansion cohort.
* Patients must have progressive disease following prior therapy. Specifically, patients must have progressed on platinum-based chemotherapy.
* At least 21 days must have elapsed from prior therapy (chemotherapy or radiation).
* Age of 18 years or older. Because no dosing or adverse event data are currently available on the use of durvalumab in combination with tremelimumab and radiation in patients <18 years of age, children are excluded from this study.
* ECOG performance status ≤1 (Karnofsky ≥60%, see Appendix A).
* Body weight of greater than 30 kg.
* Participants must have normal organ and marrow function as defined below:

  * Hgb >=9g/dl
  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin <=1.5 x normal institutional limits.

    --- This last criterion will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia [predominantly unconjugated bilirubin] in the absence of evidence of hemolysis or hepatic pathology), who will be allowed in consultation with their physician.
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal
  * Creatinine within normal institutional limits

    --- OR
  * Creatinine clearance >40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
  * Males:

    * Creatinine CL (mL/min) = Weight (kg) x (140 - Age)
    * 72 x serum creatinine (mg/dL)
  * Females:

    * Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85
    * 72 x serum creatinine (mg/dL)
* Patients must have at least one lesion not previously irradiated (and not within a previously irradiated field) for which palliative radiation to the abdomen and/or pelvis is potentially indicated and could be safely delivered at the radiation doses specified in this protocol. This lesion must not be within the CNS (brain or spinal cord), bone or liver, and must not require urgent or emergent palliative radiation given the timing of radiation specified on this protocol. Furthermore, this lesion must be located in the abdomen or pelvis and measure at least 2 cm (minimum dimension) and no greater than 6 cm (maximum dimension). Palliative radiotherapy would entail involved-field radiotherapy to a single lesion or region to encompass gross disease; whole-abdomen radiotherapy would not be permitted. Patients who received prior vaginal brachytherapy would be permitted to receive palliative pelvic radiation. In the expansion cohort at the MTD, this lesion must not be the only measurable lesion (as defined in 3.1.3) so that it is possible to determine the response rate outside of the radiation treatment field.
* The effects of durvalumab and tremelimumab on the developing human fetus are unknown. For this reason and because radiation is known to be teratogenic, evidence of post-menopausal status or negative urinary or serum pregnancy test for pre-menopausal patients is required. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced oophorectomy with last menses >1 year ago, had chemotherapy-induced menopause with >1-year interval since last menses, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
  * Women of child-bearing potential who are sexually active with a non-sterilized male partner must agree to use at least 1 method of highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 180 days after the last dose of therapy. Highly effective methods of contraception, defined as those that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, are described in section 5.5. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.

Exclusion Criteria

* Prior exposure to immune-mediated therapy, including anti-PD-1, anti-PD-L1 (including durvalumab) or anti-CTLA-4 directed therapy (including tremelimumab). Therapeutic anticancer vaccines are not included in this category. Exposure to other investigational agents may be permitted after discussion with the Study PI.
* Chemotherapy, targeted therapy, biologic or hormonal agents within 3 weeks prior to entering the study.
* Radiation therapy within 3 weeks prior to entering the study.
* Current receipt of any other investigational agents.
* Any unresolved toxicity of NCI CTCAE Grade ≥2, including electrolyte abnormalities, from previous anticancer therapy, with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Patients with untreated brain metastases, spinal cord compression, or leptomeningeal carcinomatosis are excluded from this clinical trial because of their poor prognosis, because of symptoms that may arise from inflammatory reactions, and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with brain metastases or spinal cord compression previously treated with radiation and/or surgery are allowed if local treatment was >30 days ago, most recent MRI demonstrates stability or decrease in size of all lesions, and the patient has no current neurologic symptoms related to the metastases and treatment and no requirement for corticosteroids related to the prior treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tremelimumab and durvalumab or previous toxicity attributed to durvalumab or other PD-1 or PD-L1 directed therapy that led to drug discontinuation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, interstitial lung disease, pneumonitis, active peptic ulcer disease or gastritis, active bleeding diatheses, or serious chronic gastrointestinal conditions associated with diarrhea.
* Pregnant women are excluded from this study because durvalumab and tremelimumab are immune checkpoint inhibitors with the potential for teratogenic or abortifacient effects, as is radiation therapy.
* A nursing mother unwilling to discontinue breastfeeding. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with durvalumab, tremelimumab and radiation, breastfeeding should be discontinued if the mother is treated with durvalumab, tremelimumab and radiation.
* Female patients who are pregnant or breastfeeding or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period
* HIV-positive patients are ineligible due to the risks associated with immune checkpoint blockade.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab and tremelimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as pre-medication for hypersensitivity reactions (e.g., CT scan pre-medication)
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of immunotherapy. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders. Patients without active disease in the last 5 years may be included after consultation with the study physician. This includes: inflammatory bowel disease, such as Crohn's disease or ulcerative colitis, and diverticulitis with the exception of diverticulosis; sarcoidosis syndrome, or other serious GI chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener syndrome (granulomatosis with polyangiitis); myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis; or uveitis. The following are exceptions to this criterion:

  * Vitiligo or alopecia
  * Hypothyroidism (e,g,, following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment
  * Any chronic skin condition that does not require systemic therapy
  * Celiac disease controlled by diet alone
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ)
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 consecutive electrocardiograms (EKGs) using Fridericia's Correction at baseline or before dosing. Thereafter, only 1 EKG is required during visits unless an abnormality is found and in which case, confirmation by triplicate EKGs will be needed.
* History of active primary immunodeficiency
* Known history of previous clinical diagnosis of tuberculosis
* Active infection including hepatitis B (known positive HBV surface antigen [HBsAg] result) or hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational treatment. Note: patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of investigational treatment.
* Psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational treatment or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Radiotherapy with durvalumab and tremelimumab | 8 Weeks
  Incidence of dose-limiting toxicities for each dose level or regimen

SECONDARY OUTCOMES:
Overall Response Rate | One Year
  RECIST and immune RECIST (irRC) criteria
Local Response Rate | One Year
  Response rate within the radiation field by RECIST and irRC criteria
Local Control Rate | Baseline to 6 months, 12 Months
  Tumor control within the radiation field by RECIST and irRC criteria
Abscopal Response Rate | One Year
  Abscopal response rate for measurable disease outside the radiation field by RECIST and irRC criteria
Response Duration | One Year
  Time from overall response by RECIST or irRC until time of recurrent or progressive disease
Progression Free Survival Rate | Baseline to 6 months, 12 Months
  From start of treatment to time of progression or death
Overall Survival Rate | Baseline to 6 months, 12 Months
  From start of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Martin King, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fitzgerald KJ, Konstantinopoulos P, Matulonis U, Liu J, Horowitz N, Lee E, Kolin DL, Lee L, King M. A phase I clinical trial of radiation therapy, durvalumab and tremelimumab in recurrent gynecologic cancer. Gynecol Oncol. 2025 Jun;197:51-56. doi: 10.1016/j.ygyno.2025.04.006. Epub 2025 Apr 23. PMID 40273550